CLINICAL TRIAL: NCT06574074
Title: Optimizing a Community-based Intervention to Improve Help-seeking for Depression Care in Morang District of Nepal
Brief Title: Improving Help-seeking for Depression Care in Nepal
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Transcultural Psychosocial Organization Nepal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Health Services Research
Other Study IDs: WTMOST
Record Dates: First submitted 2024-08-04; First posted 2024-08-27 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Help-Seeking Behavior; Depression
Keywords: Depression; Help-seeking behaviour; Demand side barriers; Stigma; Nepal
MeSH Terms: conditions — Help-Seeking Behavior; Depression; Social Stigma

STUDY DESIGN:
Intervention Model Description: The unit of randomization will be study participants who are identified with depression by FCHVs. Each participant will be randomized into one of eight groups using a computer-generated random number.
Who Masked: Outcomes Assessor
Masking Description: Data collectors will be blinded to the allocation of the participants to different groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (8):
- Factor-1 (Other): Participants allocated to this will receive full version of the Gain Life intervention
  Interventions: Behavioral: Gain-Life (Give informAtIoN to transform Life)
- Factor-2 (Other): Participants allocated to this will receive a few components of the Gain Life intervention that include information on depression, available treatments, and stigma reduction
  Interventions: Behavioral: Gain-Life (Give informAtIoN to transform Life)
- Factor-3 (Other): Participants allocated to this will receive only a few components of Gain Life intervention including information on depression, available treatments, and life transformation experiences
  Interventions: Behavioral: Gain-Life (Give informAtIoN to transform Life)
- Factor-4 (Other): Participants allocated to this will receive only information on depression, and available treatments components of the Gain Life intervention
  Interventions: Behavioral: Gain-Life (Give informAtIoN to transform Life)
- Factor-5 (Other): Participants allocated to this will receive three components of the Gain Life intervention that include information on depression, stigma reduction and life transformation experiences
  Interventions: Behavioral: Gain-Life (Give informAtIoN to transform Life)
- Factor-6 (Other): Participants allocated to this will receive information on depression and stigma reduction components of the Gain Life intervention
  Interventions: Behavioral: Gain-Life (Give informAtIoN to transform Life)
- Factor-7 (Other): Participants allocated to this will receive a selected components of the Gain Life intervention such as information on depression, available treatments and life transformation experiences
  Interventions: Behavioral: Gain-Life (Give informAtIoN to transform Life)
- Factor-8 (Other): Participants allocated to this will receive only the information on depression component of the Gain Life intervention
  Interventions: Behavioral: Gain-Life (Give informAtIoN to transform Life)

INTERVENTIONS:
Behavioral: Gain-Life (Give informAtIoN to transform Life) — The Gain Life intervention comprises four components: (i) information about depression, (ii) awareness of available services, (iii) stigma reduction through dispelling myths and facts about depression, and (iv) a life transformation story. The first module aims to raise awareness about depression, with a particular focus on its causes, manifestations, and the potential negative consequences of untreated depression. The second component includes the types of services offered, costs, distance to service providers, and operating hours. The third component address stigma and misconceptions surrounding depression by addressing the root causes of stigma, dispelling myths, and providing accurate information about depression. The final module of the Gain Life intervention features recovery stories of individuals who have overcome depression. This module includes two 8-minute video stories of individuals who successfully recovered from depression.

SUMMARY:
Depression is a serious public health concern worldwide due to its high prevalence rate and significant emotional and financial burden on individuals, their families, and society. There is a substantial gap between the number of people in need of treatment for depression and those who actually receive it. The recent World Health Organization (WHO) World Mental Health Survey revealed that 86.3% of people with anxiety, mood, or substance disorders in lower-middle-income countries did not receive any treatment in the past 12 months. This study aims to evaluate a community-based intervention to address demand-side barriers by improving mental health literacy, dispelling myths and misconceptions about depression, changing negative attitudes towards depression care, and promoting help-seeking behavior.

DETAILED DESCRIPTION:
It is estimated that more than 300 million people worldwide are experiencing depression, which is about 4.4% of the world's population. Despite the availability of evidence-based treatment, it is reported that 86.3% of people with anxiety, mood, or substance disorders in lower-middle-income countries received no treatment in the past 12 months. Among people who receive treatment for depression, only one out of 27 persons receive minimally adequate treatment in low- and middle-income countries (LMICs). Despite being the major contributor to the overall global burden of disease, depression receives less or no health priority in many LMICs, where more than 80% of people with depression reside.

This study will take place in two municipalities in Morang district, eastern Nepal. Female Community Health Volunteers will administer the intervention to individuals identified with depression using the locally developed and validated Community Informant Detection Tool (CIDT). Participants who receive the intervention will be followed up after one month to evaluate their help-seeking behavior (primary outcome) and after three months to assess treatment adherence, a secondary objective of the study. The study will assess the effects and interactions of four intervention components (information on depression, available treatments, stigma and myths, and life transformation experiences) on the primary outcome of help-seeking behavior and secondary outcomes such as treatment adherence. The severity of depression symptoms will be assessed using the validated PHQ-9, and knowledge and attitudes toward depression will be evaluated to assess mediation effects.

ELIGIBILITY:
Inclusion Criteria:

* being an adult aged 18 or older residing in Kanepokhari Rural Municipality or Patharisanischare Municipality,
* those detected through the CIDT
* providing consent for participation
* being proficient in speaking and understanding Nepali

Exclusion Criteria:

* people with already receiving mental health services
* having severe mental illness]
* participants below the age of 18 years,
* participants outside of Kanepokhari and Pathari-sanischare Municipality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2024-07-15 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in help-seeking behaviour for depression care | In one month
  The primary outcome of this study is "change in help-seeking behavior for depression care, defined by the proportion of participants who receive treatment from a health provider".

SECONDARY OUTCOMES:
Treatment adherence for depression | In three month
  The secondary outcome of the study is "treatment adherence for depression defined by the proportion of people who continue treatment for three months".
Change in symptom severity of depression | In three month
  The secondary outcome of the study is change in symptom severity of depression assessed by patient health questionnaire (PHQ-9). The total score of PHQ9 can range from 0 to 27, with higher scores indicating greater severity of depression
Change in knowledge, attitude and perception | In three months
  The secondary outcome of this study is to measure changes in knowledge, attitudes, and perceptions related to depression using a questionnaire developed based on the intervention content. The results will be presented based on the number of correct responses (yes and no) for each item of each scale separately. Number of greater "Yes" response indicates greater knowledge in depression, and positive attitude in help-seeking.

CONTACTS AND LOCATIONS:
Locations (1):
- Transcultural Psychosocial Organization (TPO) Nepal, Kathmandu, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No
No many researchers involved in the study so the data will only be shared within the research team

REFERENCES:
- [Derived] Luitel NP, Kohrt BA, Lamichhane B, Bhardwaj A, Gautam K, Jordans MJ. Optimizing a community-based intervention to improve help-seeking for depression care: study protocol for a randomized factorial trial. Trials. 2025 Aug 16;26(1):293. doi: 10.1186/s13063-025-09014-2. PMID 40819070